CLINICAL TRIAL: NCT07095036
Title: Generating Artificial Sensory Perceptions Using Spinal Cord Stimulation
Brief Title: Sensory Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-0213; 7DP2NS136872-02 (NIH)
Record Dates: First submitted 2025-06-16; First posted 2025-07-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Pain Management; Pain, Intractable; Pain, Chronic Disease
MeSH Terms: conditions — Agnosia; Pain, Intractable; Pain; Chronic Disease | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing sensations using spinal cord stimulation (Experimental)
  Interventions: Other: Spinal cord stimulation (SCS)

INTERVENTIONS:
Other: Spinal cord stimulation (SCS) — After implantation of SCS trial leads - which is standard of care for evaluating whether SCS improves chronic pain - patients will visit clinic before the trial leads are explanted. During these visits, stimulation will be turned off and the leads will be disconnected from the clinical external pulse generator and reconnected to an external research stimulator. Patients will be seated in a chair and will interface with a touch-screen display where they will participate in a psychophysical task (a two-alternative forced-choice task). More specifically, the task will involve selecting between two options on a screen while spinal stimulation is delivered through the leads. As the patients perform the tasks, audio or video recordings will be made for future research analysis, education, or scientific communication. The research stimulator will also collect epidural signals through the stimulation leads.

SUMMARY:
The purpose of this research study is to identify sensations that can be evoked with spinal cord stimulation (SCS) and to understand how these sensations change when stimulation parameters are modified.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-85 years old
* Undergoing SCS implantation for treatment of chronic pain
* Subjects with ability to walk 10m without assistance
* Provides written consent for the study

Exclusion Criteria:

* Subjects with high risk of falling
* Refusal to participate in study
* Subjects lacking consent capacity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Threshold amplitude for sensory perception evoked by spinal stimulation | From lead implantation to lead explantation at one week
  The outcome measure will determine the threshold stimulation amplitude in microamperes required to evoke a perceivable sensory percept during spinal stimulation.
Change in amplitude to perceive a just-noticeable difference in sensory perception evoked by spinal stimulation | From lead implantation to lead explantation at one week
  The outcome measure will determine the minimum change in stimulation amplitude in microamperes required to evoke a perceivable difference in sensory percepts during spinal stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Yadav, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Ambulatory Care Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 and continuing for 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.